CLINICAL TRIAL: NCT01762761
Title: A Multicenter, Randomized, Double-Blind and Open-label Phase III Study To Compare The Efficacy And Safety Of Eltrombopag With Placebo In Chinese Chronic ITP Patients
Brief Title: Eltrombopag Phase III Study In Chinese Chronic ITP Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113765; CETB115B2301 (Other: Novartis)
Record Dates: First submitted 2012-12-19; First posted 2013-01-08 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic and Hepatitis C
Keywords: eltrombopag; TPO-R agonist; Chronic ITP; ETB115; Chinese chronic ITP patients
MeSH Terms: conditions — Purpura; Hepatitis C | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eltrombopag (ETB115) (Experimental): Thrombopoietin- receptor (TPO-R) agonist
  Interventions: Drug: eltrombopag
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: eltrombopag — TPO-R agonist
  Other Names: ETB115
  Arms: Eltrombopag (ETB115)
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
This randomized, double-blind and open-label phase III study aimed to determine the efficacy, tolerance and safety of eltrombopag in Chinese chronic primary immune thrombocytopenia (ITP) adult subjects. This study was be conducted in Chinese adult chronic ITP subjects who had not responded to or had relapsed after previous treatment of ITP, including first line therapy and /or splenectomy.

The primary objective of this study was to determine the efficacy of oral eltrombopag as a thrombopoietic agent treating previously treated chronic Chinese ITP patients compared to placebo. The secondary objective was to assess the safety and tolerability of eltrombopag when administered for 6 weeks to previously treated adult chronic ITP patients compared with placebo. In addition, the long-term efficacy and safety of eltrombopag treatment was also evaluated in the 24-week extension open-label phase after the double-blind phase as one of other study objectives. If the subject benefited from the eltrombopag treatment based on the investigator's discretion, the subject could continue on eltrombopag treatment until the commercial launch of eltrombopag in China. Furthermore, to understand the pharmacokinetics (PK) profile of eltrombopag and to explore the relationship between the PK and pharmacodynamics (PD) (platelet response), a PK/PD analysis was embedded in this phase III study and conducted in the same patient population who participated this phase III study.

DETAILED DESCRIPTION:
This randomized, double-blind and open-label phase III study aimed to determine the efficacy, tolerance and safety of eltrombopag in Chinese chronic primary immune thrombocytopenia (ITP) adult subjects. This study was conducted in Chinese adult chronic ITP subjects who had not responded to or had relapsed after previous treatment for ITP, including first line therapy and /or splenectomy.

The primary objective of this study was to determine the efficacy of oral eltrombopag as a thrombopoietic agent treating previously treated chronic Chinese ITP patients compared to placebo. The secondary objective was to assess the safety and tolerability of eltrombopag when administered for 6 weeks to previously treated adult chronic ITP patients compared to placebo. In addition, the long-term efficacy and safety of eltrombopag treatment was also evaluated in the 24-week extension open-label phase after the double-blind phase as one of other study objectives. If the subject benefited from the eltrombopag treatment based on the investigator's discretion, the subject could continue the eltrombopag treatment until the commercial launch of eltrombopag in China. Furthermore, to understand the pharmacokinetics (PK) profile of eltrombopag and to explore the relationship between the PK and pharmacodynamics (PD) (platelet response), a PK/PD analysis was embedded in this phase III study and conducted in the same patient population who participated this phase III study.

155 eligible subjects were randomized to either eltrombopag or matching placebo treatment in 2:1 ratio in stage 1 (the 8-week double blind stage). Randomization for stage 1 was stratified by splenectomy status (Yes/No), use of concomitant maintenance ITP therapy (Yes/No) and baseline platelet count (no more than 15×109/L, or >15×109/L). This study include 3 stages. The stage 1 was an 8-week double-blind, randomized, placebo-controlled treatment period. Following completion of Stage 1 and after completing the data cleanup of the initial 6 weeks, the investigator was be un-blinded to treatment assignment on an individual subject basis to enable appropriate starting dose selection for stage 2, a 24-week open-label treatment period. PK sampling and assessments occurred at the Week 2 visit during stage 2 of the study, when all subjects were receiving eltrombopag. After the completion of stage 2, subjects could continue the the eltrombopag treatment in stage 3, if he/she benefited from the continuous eltrombopag treatment based on the investigator's judgement.

The initial dose of eltrombopag administration was an oral 25 mg once daily. During the 8 weeks double-blind treatment, dose of investigational product was adjusted according to the weekly subject platelet count.

The eligible subjects who completed stage 1 (8 weeks of double-blind treatment period: the first 6 weeks data was used for primary endpoint analysis and the last 2 weeks for data cleanup period during which the blinded treatment continued) entered a voluntary open-label stage 2 (24-week open-label extension phase) in which subjects from both the eltrombopag group and placebo group had the opportunity to receive eltrombopag treatment. Subjects unwilling or unqualified (such as the subjects who met the stopping criteria) to participate in extension treatment attended follow-up visits for 4 weeks after the completion of the double-blind phase. During the open-label stage 2 phase all eligible subjects received open label eltrombopag treatment. The dose of eltrombopag was continuously adjusted according to the subject's platelet count.

Following completion of Stage 2, if the subject benefited from the eltrombopag treatment based on the investigator's discretion, the subject could voluntarily enter stage 3, during which the subject continued eltrombopag treatment until the commercial launch of eltrombopag in C

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years old.
2. Diagnosed with ITP for at least 12 months prior to screening, and have a platelet count of <30 X109/L on Day 1 (or within 48 hours prior to dosing on Day 1).
3. Patients who have no response or relapsed after splenectomy. Or patients who have not been splenectomised and have either not responded to one or more prior therapies (except splenectomy), or who have relapsed prior therapy.
4. Previous therapy for ITP including rescue must have been completed at least 2 weeks prior to randomization.
5. Subjects treated with maintenance immunosuppressive therapy must be receiving a dose that has been stable for at least 1 month.
6. No pre-existing cardiac disease within the last 3 months. No arrhythmia known to increase the risk of thrombolic events (e.g. atrial fibrillation), or patients with a Corrected QT interval (QTc) >450msec or QTc >480 for patients with a Bundle Branch Block.
7. No history of clotting disorder, other than ITP.
8. A complete blood count (CBC), within the reference range, with the following exceptions:

   * Platelets <30×109/L on Day 1 (or within 48hours of Day 1) is required for inclusion,
   * Hemoglobin: females and males 10.0 g/dl are eligible for inclusion,
   * Absolute neutrophil count (ANC) ≥1500/µL (1.5×109/L) is required for inclusion
9. Blood chemistry test result no exceed normal by more than 20%. Total albumin must not be below the lower limit of normal (LLN) by more than 10%.
10. Subject is non-childbearing potential of childbearing potential and use acceptable methods of contraception from two weeks prior to administration of study medication, throughout the study, and 28 days after completion or premature discontinuation from the study.

Exclusion Criteria:

1. Patients with any prior history of arterial or venous thrombosis, AND ≥ two of the following risk factors: hormone replacement therapy, systemic contraception (containing estrogen), smoking, diabetes, hypercholesterolemia, medication for hypertension, cancer, hereditary thrombophilic disorders (e.g., Factor V Leiden, ATIII deficiency, antiphospholipid syndrome, etc).
2. Any clinically relevant abnormality, other than ITP,which in the opinion of the investigator makes the subject unsuitable for participation in the study.
3. Female subjects who are nursing or pregnant at screening or pre-dose on Day 1.
4. History of alcohol/drug abuse or dependence within 12 months of the study.
5. Treatment with thrombopoietin or an investigational drug within 30 days or five half-lives (whichever is longer) preceding the first dose of study medication.
6. Subjects who have previously received eltrombopag or any other thrombopoietin receptor agonist.
7. Subject has consumed aspirin, aspirin-containing compounds, salicylates, anticoagulants, quinine or non-steroidal anti-inflammatories (NSAIDs) for >3 consecutive days within 2 weeks of the study start and until the end of the study.
8. Consumption of any herbal or dietary supplements, excluding vitamin or mineral supplements, within 1 week of the study start.
9. History of platelet aggregation that prevents reliable measurement of platelet counts.
10. An abnormality in bone marrow examination result, other than ITP, identified on the screening examination, which in the opinion of the investigator makes the subject unsuitable for participation in the study (e.g. ≥MF-2 according to EU consensus scale [Thiele, 2005]) or suggests another primary diagnosis (e.g. Thrombocytopenia is secondary to another disease).
11. Any laboratory or clinical evidence for HIV infection.
12. Any clinical history for hepatitis C infection; chronic hepatitis B infection; or any evidence for active hepatitis at the time of subject screening. Laboratory test shows positive serology for Hepatitis C or Hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HB DNA test will be performed and if positive the subject will be excluded.
13. Patients expected to require rescue on Day 1 of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2013-02-18 (Actual); Primary Completion 2014-06-05 (Actual); Study Completion 2018-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- China (13):
  - Novartis Investigative Site, Fuzhou, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Zhongshan, Guangdong
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Jianan, Shandong
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chengdu
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Liu X, Hou M, Li J, Jin J, Huang M, Yu Z, Xu X, Zhang X, Yang R. Efficacy and safety of eltrombopag in Chinese patients with chronic immune thrombocytopenia: stage 2 results from a multicenter phase III study. Platelets. 2022 Jan 2;33(1):82-88. doi: 10.1080/09537104.2020.1847267. Epub 2020 Nov 29. PMID 33251910

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study includes three stages: 8-week double-blind stage (Stage 1), 24-week open-label stage (Stage 2) and prolonged open-label stage (Stage 3) with voluntary participation until eltrombopag became commercially available in China. Final Results for this study are presented in this report.
Pre-assignment Details: Participants diagnosed with primary immune thrombocytopenia (ITP) for at least 12 months prior to randomization, platelet count of <30×10^9/Liter (L) within 48 hours (hrs) prior to Day 1; no response or relapsed after splenectomy or if not splenectomised and either not responded to prior therapies or relapsed to prior therapy were enrolled.
Groups:
- Placebo: Participants initially received placebo QD. Based on weekly platelet counts, the dose of placebo was adjusted to maintain platelet counts between 50×10^9/L and 250×10^9/L for a period of 8 weeks.
- Eltrombopag: Participants initially received eltrombopag 25 milligrams (mg) QD. Based on weekly platelet counts, the dose of eltrombopag was adjusted to maintain platelet counts between 50×10^9/L and 250×10^9/L for a period of 8 weeks.
Period: Overall Study
Arm/Group | Placebo | Eltrombopag
Started | 51 | 104
Completed | 12 | 39
Not Completed | 39 | 65
Not completed — Adverse Event | 15 | 17
Not completed — Lack of Efficacy | 9 | 25
Not completed — Protocol Violation | 1 | 1
Not completed — Study closed/terminated | 0 | 2
Not completed — Lost to Follow-up | 3 | 6
Not completed — Physician Decision | 4 | 6
Not completed — Withdrawal by Subject | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Eltrombopag: Participants initially received eltrombopag 25 mg QD. Based on weekly platelet counts, the dose of eltrombopag was adjusted to maintain platelet counts between 50×10^9/L and 250×10^9/L for a period of 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Eltrombopag | Total
Number analyzed (Participants) | 51 | 104 | 155
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.3 (12.83) | 44.7 (15.91) | 43.6 (15.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 77 | 117
  Male | 11 | 27 | 38
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - East Asian Heritage | 51 | 104 | 155

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Responders) Achieving a Platelet Count >=50×10^9/L After the First 6 Weeks of Stage 1
Description: The number of participants (responders) with platelet count >=50x10^9/L after 6 weeks of Stage 1 were compared between treatments using a logistic regression model adjusted for use of primary immune thrombocytopenia (ITP) medication at Baseline (yes/no), splenectomy (yes/no), Baseline platelet count <=15×10^9/L (yes/no) and treatment. Complete blood count including platelet count was done at Week 1, Week 2, Week 3, Week 4, Week 5 and Week 6. Primary Analysis Data Set: a participant who withdrawals from Stage 1 or is emergently unblinded was classified as a negative response from the time of withdrawal or unblinding date and for all subsequent visits. In the event of a participant dying, information for all subsequent assessments would be considered missing. All intermittent missing data (apart from withdrawals) will be treated as missing.
Time Frame: From the start of study treatment (Day 1) up to the end of Week 6 of Stage 1
Population: Intent-to-Treat (ITT) Population: all randomized participants who received at least one dose of study medication and with at least one platelet count post-Baseline in Stage 1.
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 50 | 104
Participants | 3 | 60
Statistical Analysis 1: Comparison: Placebo vs Eltrombopag; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 26.08, 95% CI 2-sided [7.29 to 93.26]

2. Secondary Outcome: Number of Participants Achieving a Platelet Count >=50×10^9/L at Least Once During the First 6 Weeks of Stage 1
Description: The number of participants (responders) with platelet count >=50×10^9/L at least once during the first 6 weeks of Stage 1 were compared between treatments using a logistic regression model adjusted for use of ITP medication at Baseline (yes/no), splenectomy (yes/no), Baseline platelet count <=15×10^9/L (yes/no) and treatment. Complete blood count including platelet count was done at Week 1, Week 2, Week 3, Week 4, Week 5 and Week 6.
Time Frame: From the start of study treatment (Day 1) up to the end of Week 6 of Stage 1
Population: ITT Population: all randomized participants who received at least one dose of study medication and with at least one platelet count post-Baseline in Stage 1.
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 50 | 104
Participants | 9 | 80
Statistical Analysis 1: Comparison: Placebo vs Eltrombopag; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 23.80, 95% CI 2-sided [8.54 to 66.33]

3. Secondary Outcome: Number of Participants Achieving a Platelet Count >=30×10^9/L and at Least 2 Times the Baseline Platelet Count at Least Once During the 6 Weeks of Stage 1, the Whole Stage 2 and the Whole Stage 3
Description: The number of participants achieving a platelet count >=30×10^9/L and at least 2 times the Baseline platelet count at least once during the first 6 weeks of Stage 1 were analyzed. The Baseline platelet count is defined as the platelet count taken on Day 1 of the study or within 48 hours prior to the first dose of investigational product. Logistic regression analysis was adjusted for use of ITP medication at Baseline (yes/no), splenectomy (yes/no), Baseline platelet count <=15×10^9/L (yes/no) and treatment. Complete blood count including platelet count was done at Week 1, Week 2, Week 3, Week 4, Week 5 and Week 6.
Time Frame: From the start of study treatment (Day 1) up to the end of Stage 3
Population: ITT Population: was comprised of all rand. participats who received at least 1 dose of study medication & with at least 1 platelet count post-baseline (BL) in stages 1, 2 & 3. 1 part. did not have a BL platelet count as platelet count not collected on Day 1 or within 48 hours prior to the 1st dose of investig. product; this part. was not evaluable
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 50 | 103
Participants
  Stage 1 (during the first 6 weeks) | 18 | 84
  Stage 2 (during 24 weeks): number analyzed (Participants) | 50 | 99
  Stage 2 (during 24 weeks) | 45 | 81
  Stage 3: number analyzed (Participants) | 41 | 79
  Stage 3 | 36 | 72
Statistical Analysis 1: Comparison: Placebo vs Eltrombopag; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 8.52, 95% CI 2-sided [3.84 to 18.94]

4. Secondary Outcome: Number of Participants With Bleeding as Assessed Using the World Health Organization (WHO) Bleeding Scale
Description: The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss. The WHO Bleeding Scale were dichotomized to indicate no bleeding vs bleeding, i.e. 0=grade 0 and 1=grades 1, 2, 3 or 4. Generalized linear mixed model was applied with a Logit canonical link function for repeated binary data, allowing for Baseline dichotomized WHO bleeding grade, use of ITP medication at Baseline (yes/no), splenectomy (yes/no), Baseline platelet count <=15×10^9/L (yes/no) and treatment as fixed effects, and the participant was treated as a random effect. Bleeding incidences were recorded at Screening, Week 1, Week 2, Week 3, Week 4, Week 5 and Week 6 for Stage 1, Baseline, Weeks 4, 8, 16, 20, 24 for Stage 2; Baseline, Weeks 25, 29, 73, 97, 121, 145, 169, 193, 217, 241, 265, 284 for Stage 3. Bleeding incidences at these time points are presented.
Time Frame: From the start of study treatment (Day 1) up to the end of Stage 3
Population: ITT Population: was comprised of all rand. participats who received at least 1 dose of study medication & with at least 1 platelet count post-baseline (BL) in stages 1, 2 & 3.
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 50 | 104
Participants
  Stage 1: Baseline | 36 | 68
  Stage 1: Week 1: number analyzed (Participants) | 50 | 102
  Stage 1: Week 1 | 30 | 43
  Stage 1: Week 2: number analyzed (Participants) | 49 | 103
  Stage 1: Week 2 | 27 | 32
  Stage 1: Week 3: number analyzed (Participants) | 49 | 100
  Stage 1: Week 3 | 26 | 29
  Stage 1: Week 4: number analyzed (Participants) | 50 | 102
  Stage 1: Week 4 | 24 | 23
  Stage 1: Week 5: number analyzed (Participants) | 47 | 100
  Stage 1: Week 5 | 19 | 24
  Stage 1: Week 6: number analyzed (Participants) | 46 | 98
  Stage 1: Week 6 | 17 | 17
  Stage 2: Baseline: number analyzed (Participants) | 50 | 100
  Stage 2: Baseline | 22 | 64
  Stage 2: Week 4: number analyzed (Participants) | 40 | 28
  Stage 2: Week 4 | 8 | 7
  Stage 2: Week 8: number analyzed (Participants) | 37 | 63
  Stage 2: Week 8 | 6 | 12
  Stage 2: Week 16: number analyzed (Participants) | 33 | 52
  Stage 2: Week 16 | 5 | 8
  Stage 2: Week 20: number analyzed (Participants) | 7 | 14
  Stage 2: Week 20 | 3 | 1
  Stage 2: Week 24: number analyzed (Participants) | 33 | 61
  Stage 2: Week 24 | 3 | 6
  Stage 3: Baseline: number analyzed (Participants) | 41 | 79
  Stage 3: Baseline | 16 | 49
  Stage 3: Week 25: number analyzed (Participants) | 15 | 19
  Stage 3: Week 25 | 14 | 19
  Stage 3: Week 29: number analyzed (Participants) | 7 | 6
  Stage 3: Week 29 | 1 | 1
  Stage 3: Week 73: number analyzed (Participants) | 9 | 15
  Stage 3: Week 73 | 1 | 3
  Stage 3: Week 97: number analyzed (Participants) | 5 | 17
  Stage 3: Week 97 | 1 | 1
  Stage 3: Week 121: number analyzed (Participants) | 2 | 14
  Stage 3: Week 121 | 1 | 0
  Stage 3: Week 145: number analyzed (Participants) | 2 | 10
  Stage 3: Week 145 | 0 | 1
  Stage 3: Week 169: number analyzed (Participants) | 5 | 5
  Stage 3: Week 169 | 1 | 0
  Stage 3: Week 193: number analyzed (Participants) | 3 | 5
  Stage 3: Week 193 | 0 | 0
  Stage 3: Week 217: number analyzed (Participants) | 3 | 7
  Stage 3: Week 217 | 2 | 2
  Stage 3: Week 241: number analyzed (Participants) | 0 | 5
  Stage 3: Week 241 |  | 0
  Stage 3: Week 265: number analyzed (Participants) | 0 | 1
  Stage 3: Week 265 |  | 0
  Stage 3: Week 286: number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Eltrombopag; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Odds Ratio (OR) = 0.28, 95% CI 2-sided [0.13 to 0.59]

5. Secondary Outcome: Number of Participants With Clinically Significant Bleeding as Assessed Using the World Health Organization (WHO) Bleeding Scale
Description: The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss. The WHO Bleeding Scale grades were dichotomized into the following categories: no clinically significant bleeding = Grade 0 to 1; clinically significant bleeding = Grade 2 to 4. Generalized linear mixed model with a Logit canonical link function for repeated binary data, allowing for Baseline dichotomized WHO bleeding grade, use of ITP medication at Baseline (yes/no), splenectomy (yes/no), Baseline platelet count <=15×10^9/L (yes/no) and treatment as fixed effects, and the participant was treated as a random effect.
Time Frame: From the start of study treatment (Day 1) up to the end of Stage 3
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 50 | 104
Participants
  Stage 1: Baseline | 5 | 14
  Stage 1:Week 1: number analyzed (Participants) | 50 | 102
  Stage 1:Week 1 | 5 | 12
  Stage 1: Week 2: number analyzed (Participants) | 49 | 103
  Stage 1: Week 2 | 4 | 13
  Stage 1: Week 3: number analyzed (Participants) | 49 | 100
  Stage 1: Week 3 | 6 | 11
  Stage 1: Week 4: number analyzed (Participants) | 50 | 102
  Stage 1: Week 4 | 5 | 7
  Stage 1: Week 5: number analyzed (Participants) | 47 | 100
  Stage 1: Week 5 | 2 | 8
  Stage 1: Week 6: number analyzed (Participants) | 46 | 98
  Stage 1: Week 6 | 4 | 6
  Stage 2: Baseline: number analyzed (Participants) | 50 | 100
  Stage 2: Baseline | 3 | 13
  Stage 2: Week 4: number analyzed (Participants) | 40 | 28
  Stage 2: Week 4 | 1 | 0
  Stage 2: Week 8: number analyzed (Participants) | 37 | 63
  Stage 2: Week 8 | 0 | 1
  Stage 2: Week 16: number analyzed (Participants) | 33 | 52
  Stage 2: Week 16 | 1 | 1
  Stage 2: Week 20: number analyzed (Participants) | 7 | 7
  Stage 2: Week 20 | 1 | 0
  Stage 2: Week 24: number analyzed (Participants) | 33 | 61
  Stage 2: Week 24 | 0 | 0
  Stage 3: Baseline: number analyzed (Participants) | 41 | 79
  Stage 3: Baseline | 1 | 9
  Stage 3: Week 25: number analyzed (Participants) | 15 | 19
  Stage 3: Week 25 | 1 | 0
  Stage 3: Week 29: number analyzed (Participants) | 7 | 6
  Stage 3: Week 29 | 1 | 0
  Stage 3: Week 73: number analyzed (Participants) | 9 | 15
  Stage 3: Week 73 | 0 | 0
  Stage 3: Week 97: number analyzed (Participants) | 5 | 17
  Stage 3: Week 97 | 0 | 0
  Stage 3: Week 121: number analyzed (Participants) | 2 | 14
  Stage 3: Week 121 | 0 | 0
  Stage 3: Week 145: number analyzed (Participants) | 0 | 2
  Stage 3: Week 145 |  | 0
  Stage 3: Week 169: number analyzed (Participants) | 5 | 5
  Stage 3: Week 169 | 0 | 0
  Stage 3: Week 193: number analyzed (Participants) | 3 | 5
  Stage 3: Week 193 | 0 | 0
  Stage 3: Week 217: number analyzed (Participants) | 3 | 7
  Stage 3: Week 217 | 0 | 0
  Stage 3: Week 241: number analyzed (Participants) | 0 | 5
  Stage 3: Week 241 |  | 0
  Stage 3: Week 265: number analyzed (Participants) | 0 | 1
  Stage 3: Week 265 |  | 0
  Stage 3: Week 286: number analyzed (Participants) | 1 | 0
  Stage 3: Week 286 | 0 |
Statistical Analysis 1: Comparison: Placebo vs Eltrombopag; Test type: Superiority or Other; p = 0.306, Mixed Models Analysis; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.21 to 1.64]

6. Secondary Outcome: Time to Response
Description: Time to response is defined as time from the startin of treatment to the first time of achieving a platelet count >=50x10^9/L during the first 6 weeks of Stage 1. Time to response is summarized using Kaplan-Meier estimates and compared between treatment groups using a stratified log-rank test, stratifying for the use of ITP medication at Baseline (yes/no), splenectomy (yes/no), Baseline platelet count <=15x10^9/L (yes/no). The pike estimator of the treatment hazard ratio is based on the stratified log-rank test. Complete blood count including platelet count was done at Week 1, Week 2, Week 3, Week 4, Week 5 and Week 6.
Time Frame: From the start of study treatment (Day 1) up to the end of Week 6 of Stage 1
Population: ITT Population: was comprised of all randomized participants who received at least 1 dose of study medication & with at least 1 platelet count post-baseline in Stage 1. Only those participants with a response were analyzed.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 50 | 104
Weeks | NA [NA to NA] — The analysis was limited to only par. with a response (3 responders out of the 50 par. in the placebo group). Due to low event incidence observed in placebo group, the median time and the CI could not be calculated from the Kaplan-Meier estimates. | 3.14 [3.00 to 4.14]
Statistical Analysis 1: Comparison: Placebo vs Eltrombopag; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 6.12, 95% CI 2-sided [4.01 to 9.34]

7. Secondary Outcome: Number of Participants Who Required Protocol-defined Rescue Treatment During the First 6 Weeks of Stage 1, Whole Stages 2 & 3
Description: Rescue treatment is defined as either a new ITP medication, an increase in dose of concomitant ITP medication from Baseline, a platelet transfusion, or a splenectomy. Logistic regression analysis was adjusted for use of ITP medication at Baseline (yes/no), splenectomy (yes/no), Baseline platelet count <=15x10^9/L (yes/no) and treatment.
Time Frame: From the start of study treatment (Day 1) up to the end of Stage 3
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 50 | 104
Participants
  Stage 1 (first 6 weeks) | 17 | 9
  Stage 2: number analyzed (Participants) | 50 | 100
  Stage 2 | 16 | 14
  Stage 3: number analyzed (Participants) | 41 | 79
  Stage 3 | 13 | 21
Statistical Analysis 1: Comparison: Placebo vs Eltrombopag; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.13, 95% CI 2-sided [0.05 to 0.37]

8. Secondary Outcome: Number of Participants With a Platelet Count >=50×10^9/L During at Least 75% of Their Platelet Count Assessments
Description: The number of participants with a platelet count >=50×10^9/L during at least 75% of their platelet count assessments was analyzed up to the end of Week 6 of Stage 1. Logistic regression analysis was adjusted for use of ITP medication at Baseline (yes/no), splenectomy (yes/no), Baseline platelet count <=15x10^9/L (yes/no) and treatment. Complete blood count including platelet count was done at Week 1, Week 2, Week 3, Week 4, Week 5 and Week 6.
Time Frame: From the start of study treatment (Day 1) up to the end of Stage 3
Population: ITT Population: was comprised of all rand. participants who received at least 1 dose of study medication & with at least 1 platelet count post-baseline (BL) in stages 1, 2 & 3.
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 50 | 104
Participants
  Stage 1 (first 6 weeks) | 1 | 23
  Stage 2: number analyzed (Participants) | 50 | 100
  Stage 2 | 10 | 38
  Stage 3: number analyzed (Participants) | 41 | 79
  Stage 3 | 13 | 30
Statistical Analysis 1: Comparison: Placebo vs Eltrombopag; Test type: Superiority or Other; p = 0.008, Regression, Logistic; Odds Ratio (OR) = 16.54, 95% CI 2-sided [2.09 to 131.12]

9. Secondary Outcome: Total Duration of Time a Participant Had a Platelet Count >=50×10^9/L
Description: Total duration of time a participant had platelet count >=50 x 10^9/L was analyzed using the van Elteren stratified rank test with stratification factors including the use of ITP medication at Baseline (yes/no), splenectomy (yes/no) and Baseline platelet count <=15x10^9/L (yes/no). Complete blood count including platelet count was done at Week 1, Week 2, Week 3, Week 4, Week 5 and Week 6.
Time Frame: From the start of study treatment (Day 1) up to the end of Stage 3
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 50 | 104
Weeks
  Stage 1 (first 6 weeks) | 0.00 [0.00 to 5.1] | 1.79 [0.14 to 5.1]
  Stage 2: number analyzed (Participants) | 50 | 100
  Stage 2 | 4.07 [0.0 to 23.3] | 7.29 [0.0 to 24.6]
  Stage 3: number analyzed (Participants) | 41 | 79
  Stage 3 | 27.00 [0.0 to 227.4] | 43.71 [0.0 to 224.0]
Statistical Analysis 1: Comparison: Placebo vs Eltrombopag; Test type: Superiority or Other; p < 0.001, van Elteren stratified rank test

10. Secondary Outcome: Maximum Period of Time a Participant Had a Platelet Count Continuously >= 50 ×10^9/L
Description: Maximum period of time a participant had a platelet count continously >=50 x 10^9/L was analyzed using the van Elteren stratified rank test with stratification factors including the use of ITP medication at Baseline (yes/no), splenectomy (yes/no) and Baseline platelet count <=15x10^9/L (yes/no). Complete blood count including platelet count was done at Week 1, Week 2, Week 3, Week 4, Week 5 and Week 6.
Time Frame: From the start of study treatment (Day 1) up to the end of Stage 3
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 50 | 104
Weeks
  Stage 1 (first 6 weeks) | 0.00 [0.00 to 0.00] | 1.57 [0.14 to 3.07]
  Stage 2: number analyzed (Participants) | 50 | 100
  Stage 2 | 2.71 [0.0 to 23.3] | 5.00 [0.0 to 24.6]
  Stage 3: number analyzed (Participants) | 41 | 79
  Stage 3 | 16.43 [0.0 to 227.1] | 28.14 [0.0 to 227.1]
Statistical Analysis 1: Comparison: Placebo vs Eltrombopag; Test type: Superiority or Other; p < 0.001, van Elteren stratified rank test

11. Secondary Outcome: Number of Participants That Reduced or Discontinued Baseline Concomitant ITP Medications During Stage 2 and Stage 3
Description: The number of participants taking concomitant ITP medications on Day 1 of Stage 1 who had a decrease in the dose or frequency of ITP medication or stopped ITP medication at any point during Stage 2 or Stage 3 will be presented. The Baseline concomitant ITP medication for Stage 2 and Stage 3 is defined as ITP medications taken prior to the first dose of investigational product of Stage 1. This study is still ongoing and this endpoint can only be analyzed when the stage 2 and stage 3 complete.
Time Frame: From the start of Stage 2 to the end of Stage 3
Population: ITT Population: was comprised of all rand. participants who received at least 1 dose of study medication & with at least 1 platelet count post-baseline (BL) in stages 2 & 3.
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 50 | 100
Participants
  Stage 2 | 19 | 20
  Stage 3: number analyzed (Participants) | 41 | 79
  Stage 3 | 5 | 16

12. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product whether or not considered related to the medicinal product.A SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, is a congenital anomaly/birth defect or is associated with protocol specified liver injury and impaired liver function or is any protocol specific AEs.
Time Frame: From the start of study treatment (Day 1) up to the end of Week 8 of Stage 1
Population: Safety Population: all randomized participants who received at least one dose of the study treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 51 | 104
Participants
  Stage 1: Any AE | 34 | 66
  Stage 1: Any SAE | 5 | 5
  Stage 2: Any AE: number analyzed (Participants) | 50 | 100
  Stage 2: Any AE | 43 | 64
  Stage 2: Any SAE: number analyzed (Participants) | 50 | 100
  Stage 2: Any SAE | 6 | 11
  Stage 3: any AE: number analyzed (Participants) | 42 | 79
  Stage 3: any AE | 38 | 70
  Stage 3: Any SAE: number analyzed (Participants) | 42 | 79
  Stage 3: Any SAE | 11 | 21

13. Secondary Outcome: Number of Participants With the Maximum Toxicity Grade for the Indicated Clinical Chemistry Parameters
Description: Clinical chemistry parameters aspartate amino transferase (AST), alanine amino transferase (ALT), gamma glutamyl transferase (GGT), total bilirubin, albumin, alkaline phosphatase, calcium, potassium, creatinine, glucose and sodium were evaluated at Baseline, at all on therapy visits, and at Week 1, Week 2, Week 3, and Week 4 visits during the follow-up period and were summarized according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4 (NCI CTCAE V4.0): Grade 0, none; Grade 1, mild; Grade 2, moderate; Grade 3, severe or medically significant; Grade 4, life-threatening consequences; Grade 5, death related to AE. Day 1 assessment was considered as Baseline; if Day 1 was not available then Screening assessment is taken as Baseline. For creatinine, Baseline is defined as the average of Screening and Day 1 values if available and prior to first dose. Maximum post-Baseline toxicity grade included any scheduled or unscheduled post-Baseline assessment
Time Frame: From the start of study treatment (Day 1) up to the end of Week 6 of Stage 1
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 50 | 104
Participants
  AST, Grade 1 | 8 | 10
  AST, Grade 2 | 0 | 2
  AST, Grade 3 | 0 | 0
  AST, Grade 4 | 0 | 0
  AST, Grade 5 | 0 | 0
  ALT, Grade 1 | 11 | 14
  ALT, Grade 2 | 2 | 1
  ALT, Grade 3 | 1 | 1
  ALT, Grade 4 | 0 | 0
  ALT, Grade 5 | 0 | 0
  GGT,Grade 1 | 10 | 10
  GGT,Grade 2 | 2 | 2
  GGT,Grade 3 | 0 | 0
  GGT,Grade 4 | 0 | 0
  GGT,Grade 5 | 0 | 0
  Total Bilirubin, Grade 1 | 2 | 17
  Total Bilirubin, Grade 2 | 0 | 1
  Total Bilirubin, Grade 3 | 0 | 0
  Total Bilirubin, Grade 4 | 0 | 0
  Total Bilirubin, Grade 5 | 0 | 0
  Albumin, Grade 1 | 2 | 10
  Albumin, Grade 2 | 1 | 2
  Albumin, Grade 3 | 0 | 0
  Albumin, Grade 4 | 0 | 0
  Albumin, Grade 5 | 0 | 0
  Alkaline Phosphatase, Grade 1 | 1 | 8
  Alkaline Phosphatase, Grade 2 | 0 | 0
  Alkaline Phosphatase, Grade 3 | 0 | 0
  Alkaline Phosphatase, Grade 4 | 0 | 0
  Alkaline Phosphatase, Grade 5 | 0 | 0
  Calcium, Grade 1 | 4 | 16
  Calcium, Grade 2 | 5 | 13
  Calcium, Grade 3 | 0 | 0
  Calcium, Grade 4 | 0 | 0
  Calcium, Grade 5 | 0 | 0
  Potassium, Grade 1 | 25 | 25
  Potassium, Grade 2 | 0 | 1
  Potassium, Grade 3 | 1 | 7
  Potassium, Grade 4 | 0 | 0
  Potassium, Grade 5 | 0 | 0
  Creatinine, Grade 1 | 0 | 2
  Creatinine, Grade 2 | 0 | 0
  Creatinine, Grade 3 | 0 | 0
  Creatinine, Grade 4 | 0 | 1
  Creatinine, Grade 5 | 0 | 0
  Glucose, Grade 1 | 14 | 34
  Glucose, Grade 2 | 4 | 13
  Glucose, Grade 3 | 2 | 2
  Glucose, Grade 4 | 0 | 0
  Glucose, Grade 5 | 0 | 0
  Sodium, Grade 1 | 10 | 19
  Sodium, Grade 2 | 0 | 0
  Sodium, Grade 3 | 0 | 1
  Sodium, Grade 4 | 0 | 0
  Sodium, Grade 5 | 0 | 0

14. Secondary Outcome: Number of Participants With the Maximum Toxicity Grade for the Indicated Hematology Parameters
Description: Clinical hematology parameters hemoglobin, lymphocytes, platelet count, total neutrophils, white blood cell count evaluations were performed at Baseline, at all on-therapy visits, and at Week 1, Week 2, Week 3, and Week 4 visits during the follow-up period and were summarized according to the NCI CTCAE V4.0: Grade 0, none; Grade 1, mild; Grade 2, moderate; Grade 3, severe or medically significant; Grade 4, life-threatening consequences; Grade 5, death related to AE. Day 1 assessment was considered as Baseline; if Day 1 was not available then Screening assessment is taken as Baseline. Maximum post-Baseline toxicity grade included any scheduled or unscheduled post-Baseline assessment.
Time Frame: From the start of study treatment (Day 1) up to the end of Week 6 of Stage 1
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 50 | 104
Participants
  Hemoglobin, Grade 1 | 21 | 35
  Hemoglobin, Grade 2 | 1 | 11
  Hemoglobin, Grade 3 | 3 | 4
  Hemoglobin, Grade 4 | 0 | 0
  Hemoglobin, Grade 5 | 0 | 0
  Lymphocytes, Grade 1 | 0 | 2
  Lymphocytes, Grade 2 | 12 | 16
  Lymphocytes, Grade 3 | 0 | 1
  Lymphocytes, Grade 4 | 0 | 0
  Lymphocytes, Grade 5 | 0 | 0
  Platelet count, Grade 1 | 1 | 1
  Platelet count, Grade 2 | 0 | 11
  Platelet count, Grade 3 | 5 | 26
  Platelet count, Grade 4 | 44 | 66
  Platelet count, Grade 5 | 0 | 0
  Total Neutrophils, Grade 1 | 5 | 7
  Total Neutrophils, Grade 2 | 3 | 3
  Total Neutrophils, Grade 3 | 0 | 0
  Total Neutrophils, Grade 4 | 0 | 0
  Total Neutrophils, Grade 5 | 0 | 0
  White Blood Cell Count, Grade 1 | 4 | 9
  White Blood Cell Count, Grade 2 | 1 | 2
  White Blood Cell Count, Grade 3 | 0 | 0
  White Blood Cell Count, Grade 4 | 0 | 0
  White Blood Cell Count, Grade 5 | 0 | 0

15. Secondary Outcome: Change From Baseline in Systolic Blood Pressure
Description: Systolic blood pressure was measured in the sitting position at Baseline, Week 1, Week 2, Week 3, Week 4, Week 5 and Week 6. Day 1 assessment was considered as Baseline; if Day 1 was not available then the Screening assessment was considered as Baseline. Change from Baseline was calculated as the value at post-Baseline time point minus the value at Baseline.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5 and Week 6
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mm Hg)
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 51 | 104
Millimeters of mercury (mm Hg)
  Week 1: number analyzed (Participants) | 50 | 102
  Week 1 | -0.3 (8.86) | -0.7 (12.65)
  Week 2: number analyzed (Participants) | 49 | 103
  Week 2 | -2.0 (9.83) | -0.2 (14.08)
  Week 3: number analyzed (Participants) | 49 | 100
  Week 3 | 0.3 (12.61) | -1.5 (14.05)
  Week 4: number analyzed (Participants) | 50 | 102
  Week 4 | -0.2 (13.24) | -2.7 (14.37)
  Week 5: number analyzed (Participants) | 47 | 100
  Week 5 | -3.0 (12.02) | -2.8 (12.57)
  Week 6: number analyzed (Participants) | 46 | 98
  Week 6 | -1.5 (13.25) | -2.3 (13.62)

16. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure
Description: Diastolic blood pressure was measured in sitting position at Baseline, Week 1, Week 2, Week 3, Week 4, Week 5 and Week 6. Day 1 assessment was considered as Baseline; if Day 1 was not available then the Screening assessment was considered as Baseline. Change from Baseline was calculated as the value at post-Baseline time point minus the value at Baseline.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5 and Week 6
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 51 | 104
mm Hg
  Week 1: number analyzed (Participants) | 50 | 102
  Week 1 | -0.3 (6.66) | -0.5 (8.90)
  Week 2: number analyzed (Participants) | 49 | 103
  Week 2 | -1.1 (8.01) | -0.1 (10.91)
  Week 3: number analyzed (Participants) | 49 | 100
  Week 3 | -1.0 (7.16) | -1.5 (10.40)
  Week 4: number analyzed (Participants) | 50 | 102
  Week 4 | -0.9 (8.51) | -1.4 (9.57)
  Week 5: number analyzed (Participants) | 47 | 100
  Week 5 | -3.0 (8.39) | -1.8 (9.78)
  Week 6: number analyzed (Participants) | 46 | 98
  Week 6 | -2.2 (9.44) | -1.0 (9.71)

17. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was measured at Baseline, Week 1, Week 2, Week 3, Week 4, Week 5 and Week 6. Day 1 assessment was considered as Baseline; if Day 1 was not available then the Screening assessment was considered as Baseline. Change from Baseline was calculated as the value at post-Baseline time point minus the value at Baseline.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5 and Week 6
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 51 | 104
Beats per minute
  Week 1: number analyzed (Participants) | 50 | 102
  Week 1 | -0.5 (6.88) | 0.2 (8.54)
  Week 2: number analyzed (Participants) | 49 | 103
  Week 2 | -2.2 (9.23) | 0.2 (9.54)
  Week 3: number analyzed (Participants) | 49 | 100
  Week 3 | 1.6 (10.31) | 0.2 (8.79)
  Week 4: number analyzed (Participants) | 50 | 102
  Week 4 | -0.1 (7.32) | 0.8 (8.52)
  Week 5: number analyzed (Participants) | 47 | 100
  Week 5 | 0.0 (9.06) | 0.0 (7.32)
  Week 6: number analyzed (Participants) | 46 | 98
  Week 6 | -2.1 (8.55) | 0.1 (8.06)

18. Secondary Outcome: Number of Participants With the Indicated 12-lead Electrocardiogram (ECG) Finding at Baseline
Description: Resting 12-lead ECG was obtained at Baseline. Day 1 assessment was considered as Baseline; if Day 1 was not available then the Screening assessment was considered as Baseline. ECG was also obtained when there was clinical symptom that potentially related to cardiac dysfunction based on investigator's judgement.
Time Frame: Baseline
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Particpants
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 50 | 104
Particpants
  Normal | 36 | 57
  Abnormal, not clinically significant | 14 | 43
  Abnormal, clinically significant | 0 | 4

19. Secondary Outcome: Number of Participants With a Change From Baseline in Visual Acuity
Description: Visual acuity is a measure of the spatial resolution of the visual processing system. Acuity is a measure of visual performance and is unrelated to the eyeglass prescription required to correct vision. Normal visual acuity is commonly referred to as 20/20 vision. Evaluation was done for oculus sinister (OS) for the left eye, oculus dexter (OD) for the right eye. Change from Baseline was calculated as the value at post-Baseline time point minus the value at Baseline.
Time Frame: From the start of study treatment (Day 1) up to the end of Week 6 of Stage 1
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 51 | 104
Participants
  OD | 24 | 33
  OS | 22 | 35

20. Secondary Outcome: Number of Participants With the Indicated Grading of Myelofibrosis Using Bone Marrow Biopsy at Screening
Description: Bone marrow biopsy was performed at Screening and then obtained when clinically indicated. Whenever a peripheral blood smear confirmed the presence of immature or dysplastic cells, a bone marrow examination was performed. Myelofibrosis (MF) was graded from Grade MF-0 to MF-3 where MF-0=scattered linear reticulin with no intersections (cross-overs) corresponding to normal bone marrow; MF-1=loose network of reticulin with many intersections; especially in perivascular areas; MF-2=diffuse and dense increase in reticulin with extensive intersections, occasionally with only focal bundles of collagen and/or focal osteosclerosis; MF-3=diffuse and dense increase in reticulin with extensive intersections with coarse bundles of collagen, often associated with significant osteosclerosis.
Time Frame: Screening
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Eltrombopag
Number analyzed (Participants) | 51 | 102
Participants
  MF Score 0 | 38 | 83
  MF Score 1 | 13 | 19
  MF Score 2 | 0 | 0
  MF Score 3 | 0 | 0

21. Secondary Outcome: Pharmacokinetic (PK) Assessments for Eltrombopag for Apparent Volume of Distribution of Central Compartment (Vc/F), Apparent Volume of Distribution of Peripheral Compartment (Vp/F)
Description: Vc/F is apparent volume of distribution of plasma (VDP) in central compartment and Vp/F is apparent VDP in peripheral compartment. PK assessments were made with one group of serial sampling [Samples collected at pre-dose and 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 24 hr post-dose] and one group of sparse assessment [Samples collected at pre-dose, between 2 to 4 hr and 5 to 8 hr post-dose]. Pre-dose samples were collected within 2 hr prior to dosing, all other samples were collected within 10 minutes(min) for samples collected between 1 and 6 hrs and within 30 mins for samples collected at 8 and 24 hr. PK analysis was conducted using a population approach with non-linear mixed effects modeling methods. Point estimates of population PK parameters are presented.
Time Frame: From the start of study until 24 hours post-dose of Week 2 Visit of Stage 2
Population: PK Population: all participants with evaluable dosing, actual sampling time, and eltrombopag concentration data.
Measure: Geometric Mean (95% Confidence Interval); unit: Liters
Groups:
- Eltrombopag: In Stage 1, Participants were given placebo QD for 8 weeks or were initially treated with 25 mg eltrombopag. Dose of eltrombopag was adjusted to maintain platelet counts between 50×10^9/L and 250×10^9/L for period of 8 weeks based on weekly platelet counts. In Stage 2, participants who received eltrombopag in Stage 1 continued with the same dose of eltrombopag unless the platelet count warranted an adjustment. Participants who received placebo in Stage 1 started 25 mg eltrombopag once daily as the initial dose and was adjusted to maintain platelet counts between 50×10^9/L and 250×10^9/L for period of 8 weeks on based on weekly platelet counts.
Arm/Group | Eltrombopag
Number analyzed (Participants) | 148
Liters
  Vc/F | 8.80 [7.84 to 9.76]
  Vp/F | 33.6 [17.0 to 50.2]

22. Secondary Outcome: Pharmacokinetic Assessments for Eltrombopag for Apparent Clearance (CL/F), Apparent Inter-compartmental Clearance (Q/F)
Description: CL/F is defined as the apparent oral clearance from plasma and Q/F is defined as apparent intercompartmental clearance. PK assessments were made with one group of serial sampling [Samples collected at pre-dose and 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 24 hr post-dose] and one group of sparse assessment [Samples collected at pre-dose, between 2 to 4 hr and 5 to 8 hr post-dose]. Pre-dose samples were collected within 2 hr prior to dosing, all other samples were collected within 10 min for samples collected between 1 and 6 hr and within 30 min for samples collected at 8 and 24 hr. PK analysis was conducted using a population approach with non-linear mixed effects modeling methods. Point estimates of population PK parameters are presented.
Time Frame: From the start of study until 24 hours post-dose of Week 2 Visit of Stage 2
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Liters per hour(L/hr)
Arm/Group | Eltrombopag
Number analyzed (Participants) | 148
Liters per hour(L/hr)
  CL/F | 0.370 [0.336 to 0.404]
  Q/F | 0.561 [0.444 to 0.678]

23. Secondary Outcome: Pharmacokinetic Assessments for Eltrombopag for Absorption Rate Constant (Ka)
Description: Ka is defined as the absorption rate constant. PK assessments were made with one group of serial sampling [Samples collected at pre-dose and 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 24 hr post-dose] and one group of sparse assessment [Samples collected at pre-dose, between 2 to 4 hr and 5 to 8 hr post-dose]. Pre-dose samples were collected within 2 hrs prior to dosing, all other samples were collected within 10 min for samples collected between 1 and 6 hrs and within 30 mins for samples collected at 8 and 24 hr. PK analysis was conducted using a population approach with non-linear mixed effects modeling methods. Point estimates of population PK parameter is presented.
Time Frame: From the start of study until 24 hours post-dose of Week 2 Visit of Stage 2
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Per hour (1/hr)
Arm/Group | Eltrombopag
Number analyzed (Participants) | 148
Per hour (1/hr) | 1.58 [1.05 to 2.11]

24. Secondary Outcome: Pharmacokinetic Assessments for Eltrombopag for Absorption Lag Time (ALAG)
Description: Absorption lag time (ALAG) is defined as the time taken for a drug to appear in the systemic circulation following administration. PK assessments were made with one group of serial sampling [Samples collected at pre-dose and 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 24 hr post-dose] and one group of sparse assessment [Samples collected at pre-dose, between 2 to 4 hrs and 5 to 8 hrs post-dose]. Pre-dose samples were collected within 2 hrs prior to dosing, all other samples were collected within 10 min for samples collected between 1 and 6 hr and within 30 min for samples collected at 8 and 24 hr. PK analysis was conducted using a population approach with non-linear mixed effects modeling methods. Point estimates of population PK parameter is presented.
Time Frame: From the start of study until 24 hours post-dose of Week 2 Visit of Stage 2
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Hour
Arm/Group | Eltrombopag
Number analyzed (Participants) | 148
Hour | 0.855 [0.816 to 0.894]

25. Secondary Outcome: Post-hoc Estimates of Plasma Eltrombopag Area Under the Concentration-time Curve Over a Dosing Interval (AUC[0-tau]) After 50 mg Once Daily Dose of Eltrombopag
Description: AUC[0-tau] is defined as area under the concentration-time curve over a dosing interval (24 hr) of Eltrombopag atsteady-state after 50 mg once daily dose of eltrombopag. PK analysis was conducted using a population approach with non-linear mixed effects modeling methods. Post-hoc estimates of steady-state eltrombopag was determined based on the final PK model. Individual PK parameters were derived from the final PK model by an empirical Bayes estimation. Summary of steady-state AUC(0-tau) of eltrombopag is presented here.
Time Frame: From the start of study until 24 hours post-dose of Week 2 Visit of Stage 2
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram* hour per milliliter(μg.hr/mL)
Arm/Group | Eltrombopag
Number analyzed (Participants) | 148
Microgram* hour per milliliter(μg.hr/mL) | 88.8 [78.0 to 101]

26. Secondary Outcome: Post-hoc Estimates of Maximum Observed Concentration (Cmax) for Eltrombopag After 50 mg Once Daily Dose of Eltrombopag
Description: Cmax is defined as maximum observed concentration after 50 mg once daily dose of eltrombopag. PK analysis was conducted using a population approach with non-linear mixed effects modeling methods. Post-hoc estimates of steady-state eltrombopag Cmax was determined based on the final PK model. Individual PK parameters were derived from the final PK model by an empirical Bayes estimation. Summary of steady-state Cmax of eltrombopag .is presented here.
Time Frame: From the start of study until 24 hours post-dose of Week 2 Visit of Stage 2
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Nanogram/ Milliliter (ng/mL)
Arm/Group | Eltrombopag
Number analyzed (Participants) | 148
Nanogram/ Milliliter (ng/mL) | 6916 [6205 to 7708]

27. Secondary Outcome: Percentage of Participants Estimated as Responders to Eltrombopag by the Pharmacokinetic/ Pharmacodynamic Model
Description: Responders are participants whose SLOP estimates are larger than zero. The Pharmacokinetic/ Pharmacodynamic relationship between eltrombopag concentrations and the platelet response was described by a four-compartment life span model, representing one precursor production compartment, two transit/maturation compartments and one blood platelet compartment.
Time Frame: From the start of study until 24 hours post-dose of Week 2 Visit of Stage 2
Population: PK/PD Population: all participants with evaluable dosing, actual sampling time, and platelet count data.
Measure: Number; unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 147
Percentage of participants | 89

28. Secondary Outcome: Pharmacodynamic Parameter-Linear Proportionality Constant of Drug Effect (SLOP): the Proportional Increase of Platelet Production Rate With Each 1-μg/mL Increase in Eltrombopag Plasma Concentration
Description: The Pharmacokinetic/ Pharmacodynamic relationship between eltrombopag concentrations and the platelet response was described by a four-compartment life span model, representing one precursor production compartment, two transit/maturation compartments and one blood platelet compartment.
Time Frame: From the start of study until 24 hours post-dose of Week 2 Visit of Stage 2
Population: PK/PD Population
Measure: Geometric Mean (95% Confidence Interval); unit: Milliliter/microgram
Arm/Group | Eltrombopag
Number analyzed (Participants) | 147
Milliliter/microgram | 0.860 [0.639 to 1.08]

29. Secondary Outcome: Pharmacodynamic Parameter- Production Rate of Platelet Precursors (KIN)
Description: The Pharmacokinetic/ Pharmacodynamic relationship between eltrombopag concentrations and the platelet response was described by a four-compartment life span model, representing one precursor production compartment, two transit/maturation compartments and one blood platelet compartment. The estimate of KIN was fixed to 1.43x10^9/L.hr.
Time Frame: From the start of study until 24 hours post-dose of Week 2 Visit of Stage 2
Population: PK/PD Population
Measure: Number; unit: 1 x 10^9/L.hr
Arm/Group | Eltrombopag
Number analyzed (Participants) | 147
1 x 10^9/L.hr | 1.43

30. Secondary Outcome: Pharmacodynamic Parameter-Maturation Rate of Platelet Precursors (KOUT)
Description: The Pharmacokinetic/ Pharmacodynamic relationship between eltrombopag concentrations and the platelet response was described by a four-compartment life span model, representing one precursor production compartment, two transit/maturation compartments and one blood platelet compartment. The estimate of KOUT was fixed to 0.0253 /hr.
Time Frame: From the start of study until 24 hours post-dose of Week 2 Visit of Stage 2
Population: PK/PD Population
Measure: Number; unit: 1/ hr
Arm/Group | Eltrombopag
Number analyzed (Participants) | 147
1/ hr | 0.0253

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) timeframe: Adverse events were collected from study start (form first dose of study treatment) until end of study treatment plus 30 days post-treatment, up to a maximum duration of approx. 70 months.
Description: Adverse Event (AE): Any sign or symptom that occurs during the study treatment plus the 30 days post treatment
Arm/Group | Placebo | Eltrombopag
All-Cause Mortality (participants affected / at risk) | 3/51 | 0/104
Serious Adverse Events (participants affected / at risk) | 17/51 | 33/104
Other Adverse Events (participants affected / at risk) | 48/51 | 90/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | Eltrombopag (N=104)
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 3
THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 0
THYROIDITIS SUBACUTE (Endocrine disorders) | 0 | 1
CATARACT (Eye disorders) | 1 | 4
CATARACT SUBCAPSULAR (Eye disorders) | 0 | 1
LENTICULAR OPACITIES (Eye disorders) | 1 | 0
RETINOPATHY (Eye disorders) | 0 | 1
GASTRIC POLYPS (Gastrointestinal disorders) | 0 | 1
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1
HIATUS HERNIA (Gastrointestinal disorders) | 0 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
INTUSSUSCEPTION (Gastrointestinal disorders) | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
CHEST DISCOMFORT (General disorders) | 0 | 1
DEATH (General disorders) | 2 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1
GASTROENTERITIS (Infections and infestations) | 1 | 0
HERPES ZOSTER (Infections and infestations) | 1 | 0
LUNG INFECTION (Infections and infestations) | 0 | 2
RECTAL ABSCESS (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FRACTURED COCCYX (Injury, poisoning and procedural complications) | 0 | 1
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 0 | 1
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
BILIRUBIN CONJUGATED INCREASED (Investigations) | 0 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 1
HEPATIC ENZYME INCREASED (Investigations) | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 4 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 1
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
SJOGREN'S SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 0 | 1
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SEMINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BRAIN STEM HAEMORRHAGE (Nervous system disorders) | 1 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 1 | 4
CEREBROVASCULAR INSUFFICIENCY (Nervous system disorders) | 0 | 1
NEURALGIA (Nervous system disorders) | 0 | 1
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 | 0
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 2
CALCULUS URINARY (Renal and urinary disorders) | 1 | 0
GYNAECOMASTIA (Reproductive system and breast disorders) | 0 | 1
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 1
OVARIAN CYST RUPTURED (Reproductive system and breast disorders) | 0 | 1
ABORTION INDUCED (Surgical and medical procedures) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
NECROSIS ISCHAEMIC (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | Eltrombopag (N=104)
ANAEMIA (Blood and lymphatic system disorders) | 9 | 17
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 2 | 8
VISION BLURRED (Eye disorders) | 3 | 7
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 7
DIARRHOEA (Gastrointestinal disorders) | 8 | 11
GINGIVAL BLEEDING (Gastrointestinal disorders) | 4 | 0
TOOTHACHE (Gastrointestinal disorders) | 1 | 7
CHEST DISCOMFORT (General disorders) | 3 | 2
FATIGUE (General disorders) | 4 | 5
OEDEMA PERIPHERAL (General disorders) | 4 | 3
PYREXIA (General disorders) | 4 | 2
GINGIVITIS (Infections and infestations) | 2 | 7
NASOPHARYNGITIS (Infections and infestations) | 21 | 28
PHARYNGITIS (Infections and infestations) | 5 | 10
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 13 | 39
URINARY TRACT INFECTION (Infections and infestations) | 13 | 19
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 19 | 26
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 18 | 22
BILIRUBIN CONJUGATED INCREASED (Investigations) | 4 | 11
BLOOD BILIRUBIN INCREASED (Investigations) | 9 | 19
BLOOD BILIRUBIN UNCONJUGATED INCREASED (Investigations) | 10 | 10
BLOOD CREATININE INCREASED (Investigations) | 4 | 2
BLOOD GLUCOSE INCREASED (Investigations) | 2 | 9
BLOOD UREA INCREASED (Investigations) | 2 | 6
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 8 | 12
NEUTROPHIL COUNT DECREASED (Investigations) | 3 | 1
NEUTROPHIL COUNT INCREASED (Investigations) | 3 | 7
RETICULOCYTE COUNT INCREASED (Investigations) | 3 | 2
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 3 | 3
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 6 | 5
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 3 | 4
HYPERURICAEMIA (Metabolism and nutrition disorders) | 4 | 4
HYPOKALAEMIA (Metabolism and nutrition disorders) | 14 | 20
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 6
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 7
DIZZINESS (Nervous system disorders) | 3 | 7
HEADACHE (Nervous system disorders) | 3 | 8
PROTEINURIA (Renal and urinary disorders) | 3 | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 7
PRURITUS (Skin and subcutaneous tissue disorders) | 4 | 4
RASH (Skin and subcutaneous tissue disorders) | 7 | 7
HYPERTENSION (Vascular disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety